CLINICAL TRIAL: NCT07132554
Title: Mixing 1:1 HIIT and MICT in Early to Very Early Phase Heart Transplant (HTx) Recipients : a Retrospective Study From a 510 Patients/12 Years Prospectively-collected Database
Brief Title: Mixing 1:1 HIIT and MICT in Early to Very Early Phase HTx Recipients : a Retrospective Study From a 510 Patients/12 Years Database
Acronym: COMET-HT
Status: Completed | Type: Observational
Sponsor: Hôpital Léon Bérard (Other)
Collaborators: Groupement des Hôpitaux de l'Institut Catholique de Lille (GHICL) - France (Unknown); Centre Hospitalier Toulon (Unknown)
Responsible Party: Principal Investigator, Benjamin BERNUZ, MD, Scientific coordinator, Hôpital Léon Bérard
Other Study IDs: COMET-HT2012-2024
Record Dates: First submitted 2025-07-22; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Heart Transplant Recipients
Keywords: Exercise-based cardiac rehabilitation; VO2peak; Combine Moderate and Intense Training; Early-to-very-early phase post-HTx; Exercise capacity determinants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Combined 1:1 MICT and HIIT aerobic cardiac rehabilitation — Combining 1:1 MICT and HIIT in short (4 weeks) high-volume (32 sessions) early-to-very-early phase program post heart transplantation

SUMMARY:
Background: Exercise-based cardiac rehabilitation is recommended early to very early for heart transplant recipients (HTRs), but data on its feasibility and efficacy at this stage are lacking. Primarily, this study reports the results of an intensive program combining moderate-intensity continuous-training (MICT) and high-intensity interval-training (HIIT) in early HTRs. Secondarily, it explores the determinants of VO2peak in this population.

Methods: A single-center retrospective study of a prospectively-collected database including patients who were consecutively referred to a cardiac rehabilitation unit immediately after discharge from acute post-transplant care, between December 2012 and December 2024. Patients participated in a tailored program combining MICT and HIIT as soon as they could cycle, and performed a first cardiopulmonary exercise test (CPET1) when possible. The initial prescription included 32 planned 30-minute (±5) aerobic sessions for 4 weeks, on a standard or semi-recumbent cycle-ergometer, twice a day (4 days a week) including one session of MICT (PVT and Borg-RPE 12-14) and one session of HIIT (6-8 x 1':3'/ PAT and Borg-RPE ≥ 15), plus additional sessions (respiratory and strengthening physiotherapy, gymnastics or walking, occupational therapy). The primary outcome was improvement in exercise capacity, measured by maximal oxygen consumption (VO2peak) between CPET1 and discharge (CPET2). Secondary outcomes included feasibility criterions (exercise-related adverse events-AE, and completion rates), then clinical, biological and echocardiographic parameters influencing exercise capacity.

DETAILED DESCRIPTION:
INTRODUCTION The incidence and prevalence of heart failure (HF) are increasing globally. While its prevalence is estimated at 2% in developed countries, a similar upward trend has been observed in developing countries since the 2000s. This growing burden has led to a parallel rise in cases of advanced HF, a trend primarily driven by an aging population and improved patient survival rates. For patients with advanced HF and no contraindications, heart transplantation (HTx) remains the gold-standard treatment.

Concurrently, exercise capacity is a critical health indicator. In the general population, it is recognized as the strongest predictor of good health and survival, regardless of underlying pathologies. This importance is mirrored in heart transplant recipients (HTR), where enhanced exercise capacity is associated with improved functional status, better quality of life and lower re-hospitalization rates. Furthermore, emerging evidence suggests an inverse relationship with post-transplant mortality. For instance, a +14% increase in maximal oxygen consumption (VO2peak) has been estimated to yield a 32% reduction in mortality.

Exercise-based cardiac rehabilitation programs are the primary intervention for improving exercise capacity after HTx. Their effectiveness in increasing VO2peak was confirmed by a meta-analysis of nine randomized controlled trials (284 patients), the majority of which (n=8) utilized Moderate-Intensity Continuous Training (MICT), yielding a significant mean difference of +2.49 ml/kg/min (95% CI 1.69 to 3.49). However, these studies have limitations. With one exception from the smallest, the trials were conducted in the stable, chronic phase post-HTx (median 12 months) and exhibited significant heterogeneity in the type, volume, and intensity of aerobic exercise prescribed. Notably, despite being a major determinant of program effectiveness, patient adherence was not reported in any of these studies.

A few retrospective studies with small to medium sample sizes, more recently, the largest randomized controlled trial (n=81) to date have explored the effects of early cardiac rehabilitation. While these programs started between 2 and 3 months after HTx, few data exist on very early (≈1 month) standardized rehabilitation programs. In addition, if the ability of MICT to improve cardiorespiratory fitness (CRF) in HTx has been demonstrated, Nytroen et al. demonstrated the efficacy and safety of high-intensity interval training (HIIT) over MICT (SMD +1.8 mL/kg/min), in a long-term (9 months), high-volume (58 sessions x 25 minutes), high-intensity, good adherence, out-patient program.

Yet, recommendations still suggest starting at low intensity (≤50% VO2peak or -10% below the VO2ventilatory threshold), from the 2nd or 3rd post-operative week for the first few weeks, then increasing to MICT and then HIIT depending on tolerance, whereas HIIT should be introduced " only in the further course of clinically stable patient ". However, it may be that initial adherence to and enjoyment of exercise is a cornerstone of long-term physical activity maintenance Rodrigues, especially in the context of HF Klompstra. As described in other population, early in-center peer emulation and addressing the monotony of exercise programs seem important for improving initial management and long-term adherence.

The aim of this study is to report the feasibility and efficacy of an early to very early standardized mixed HIIT/MICT rehabilitation program in HTR implemented in routine care at our institution, as well as to explore some prognostic parameters related to early initial exercise capacity.

METHODS The study was conducted in accordance with the Declaration of Helsinki. All participants provided written informed consent for their anonymized data to be used for research purposes. The study protocol was approved by the relevant institutional review board. The datasets used and/or analysed during the current study have been submitted to the editor. Data are available from the corresponding author on reasonable request.

2.1. Objectives The primary objective of this study was to evaluate the change in exercise capacity, measured by cardiopulmonary exercise testing, in heart transplant recipients between admission (CPET1) and discharge (CPET2) from an intensive mixed HIIT/MICT rehabilitation program. The secondary objective was to conduct an exploratory analysis to identify the determinants of exercise capacity in this population.

The primary endpoint was change in VO2peak between CPET1 and CPET2. The secondary endpoints were change between all other CPET parameters, and an exploratory analysis of the clinical, biological and echocardiographic determinants of exercise capacity.

2.2. Study Design and Population This retrospective cohort study was conducted using data from a single, specialized cardiac rehabilitation center (Hôpital Léon Bérard, Hyères, France). The investigators included all HTR (n=510) admitted between December 2012 and February 2023 for early inpatient rehabilitation. All participants were referred from three French university hospital transplant centers (CHU La Timone, Marseille; CHU Edouard Herriot, Lyon; and CHU Arnaud de Villeneuve, Montpellier) immediately after their acute post-surgical phase.

2.3. Data Collection Data were sourced from a local database created for this population in December 2012. The collection process was hybrid: data from December 2012 to June 2019 were extracted retrospectively from digitized medical records, whereas data from July 2019 onward were entered prospectively by the two attending cardiologists.

2.4. General process The general procedure for all admitted patients was prescribed and managed by two cardiologists, each with over two decades of experience, while daily field management was conducted by a dedicated team of physiotherapists and adapted physical activity (APA) instructors. All training sessions took place in an open-space environment under continuous cardiac monitoring and the direct supervision of an on-site cardiologist. The program included a comprehensive baseline assessment during the first week, comprising clinical data, routine biological parameters, a resting echocardiogram, and a cardiopulmonary exercise test (CPET1), repeated at discharge during the final week (CPET2). The 4-week intervention was structured around a high-frequency aerobic training regimen, complemented by a supplemental program adjusted for patient fatigue. The primary aerobic program, for patients able to perform CPET1, followed the FITT principle: Frequency of 8 sessions per week (twice daily, 4 days/week); Intensity prescribed in a target range between the first (VT₁) and second (VT₂) ventilatory thresholds; Time of 30 ± 5 minutes per session; and Type of exercise on a standard or semi-recumbent cycle ergometer. The supplemental program consisted of respiratory physiotherapy (4 sessions/week), resistance training (2 sessions/week, progressing from 30% to 50% of 1-RM), group activities such as outdoor walking or gymnastics (2 sessions/week), and occupational therapy. For patients unable to perform the CPET1, a modified protocol was implemented, typically involving one to two daily sessions of 15 to 30 minutes of moderate-intensity continuous training (MICT), with intensity guided by a Borg RPE of 12-14 on a semi-recumbent or arm ergometer. It should be noted that the subsequent analyses described in this paper pertain specifically to the cohort of patients who completed the baseline CPET.

2.5. Patient Assessment Protocol 2.5.1 Cardiopulmonary exercise testing The primary endpoint was the change in peak oxygen uptake (VO₂peak) from baseline to discharge.

Exercise capacity was assessed using a symptom-limited, incremental cardiopulmonary exercise test (CPET) performed on a standard or semi-recumbent cycle ergometer (ERGOLINE, Geispolsheim, France; or Corival CPET, Lode B.V., Groningen, The Netherlands). Each test began with a 2-minute warm-up (0-20 W) at a target cadence of 60 ± 10 rpm. Following the warm-up, an individualized ramp protocol was initiated, chosen from one of the following to target an optimal test duration of 8 ± 2 minutes:

An increment of 5 W/min after a 1-minute stage at 7 W (Corival ergometer protocol).

An increment of 5 W/min after a 1-minute stage at 20 W. An increment of 10 W/min after a 1-minute stage at 20 W. The test was continued until volitional exhaustion, with strong verbal encouragement provided. Test termination criteria adhered to the recommendations of the American College of Sports Medicine, and a 5- to 6-minute recovery period was systematically performed. A peak respiratory exchange ratio (RER) of ≥1.15 was considered the criterion for a maximal effort.

Gas exchange and ventilatory variables were measured on a breath-by-breath basis using a metabolic cart (METASYS TR-M, Brainware, La Valette du Var, France) and averaged every 15 seconds. Continuous 12-lead electrocardiography monitored heart rate (HR), while blood pressure was measured manually every two minutes.

The following specific parameters were selected for analysis:

Peak Exercise Values: Peak oxygen uptake (VO₂peak), defined as the highest VO₂ recorded; maximal power output (Pₘₐₓ); peak heart rate (HRₚₑₐₖ); peak minute ventilation (VEₚₑₐₖ); and the peak respiratory exchange ratio (RER).

Submaximal Thresholds: Values for VO₂, power (P), and HR were determined at the first and second ventilatory thresholds (VT₁ and VT₂, respectively).

Derived and Relative Parameters: The O₂ pulse (VO₂peak / HRₚₑₐₖ) was calculated. All absolute values for VO₂, P, and HR at peak exercise and at the ventilatory thresholds were also expressed as a percentage of their age-predicted norms based on the Wasserman equations.

2.4.2 6 min walk test

2.5. Rehabilitation program All rehabilitation sessions were conducted on an inpatient basis at the Hôpital Léon Bérard. Upon admission, each patient's comprehensive rehabilitation program was prescribed by a cardiologist and individually tailored based on their physical capacity, as determined by an initial physical therapy assessment and baseline cardiopulmonary exercise test (CPET1) results. The care of all heart transplant recipients (HTR) was specifically overseen by two dedicated cardiologists. The program consisted of twice-daily training sessions (morning and afternoon), five days a week (Monday to Friday), all conducted under the direct supervision of a physical therapist or a specialized Adapted Physical Activity (APA) instructor. For safety, a cardiologist was continuously available in close proximity to the training facility. As detailed in Table 1, the multi-component intervention integrated tailored endurance and resistance training, daily respiratory physiotherapy, collective physical activities, and a multi-faceted therapeutic education curriculum. A complete description of the specific protocols, intensity targets, session frequencies, and corresponding patient profiles for each intervention is provided in Table 1.

Table 1. Comprehensive Cardiac Rehabilitation Program Component / Activity Target Patient Profile Frequency Protocol / Details Endurance: Cycling / Ergoline Patients who can perform an CPET with no contraindication to cycling. 2 sessions / day (adjusted for fatigue) Session 1 (Moderate Intensity Continuous Training): 5 min warm-up + 25-40 min at aerobic threshold (VT1), maintaining a Borg scale rating of 12-14.

Session 2 (High intensity Interval Training - HIIT): 5 min warm-up + 24-38 min. Protocol: 1 min at anaerobic threshold (VT2) followed by 3 min recovery below VT1.

Endurance: Alternative Protocol Patients with very low capacity, or who have contraindications or an aversion to standard protocols.

1-2 sessions / day Moderate Intensity Continuous training: 15-30 min on Motomed (Borg 12-14) or treadmill (low/no incline, speed set to Borg 12-14); increasing if possible to HIIT at the end of the program.

Respiratory Physiotherapy All patients.

1. session / day Performed on a therapy table. Focuses on diaphragmatic breathing and mobilizing respiratory volumes to counter the effects of sternotomy. Includes light limb strengthening (1-2 kg weights).

   Quadriceps Strengthening All patients, as soon as possible. 2-3 times / week Using a leg extension machine (3 sets of 10 reps).
   * Week 1: 30% of 1-Repetition Maximum (1RM)
   * Week 2: 40% of 1RM
   * Week 3: 50% of 1RM

   Autonomy Rehabilitation Patients with a significant loss of autonomy. As needed Physiotherapy/Occupational therapy sessions for verticalization, transfers (e.g., wheelchair to table), and progressive rehabilitation for walking and climbing stairs.

   Individualized care following a functional neuromuscular and cognitive assessment.

   Group Gymnastics All patients, grouped by physical capacity.
2. session / week
3. Levels:

   * Low Intensity: Seated exercises, transfer practice, balance.
   * Moderate Intensity: Standing exercises, postural work, avoiding sternal stress.
   * High Intensity: Standing exercises at a high pace with more repetitions. Group Walk All patients capable of walking on uneven ground.

2 session / week

Outdoor walk in the hospital park, split into two groups:

* Moderate: 1.1 km in 25 min (~2.6 km/h).
* Intense: 2.3 km in 34 min (~4.2 km/h).

Therapeutic Education: Medication All cardiac transplant patients. Scheduled workshop A group session on medication management, led by pharmacists. Therapeutic Education: Diet & Nutrition All cardiac transplant patients. Throughout the stay Led by dietitians, program includes an initial assessment, an educational workshop, and a final assessment.

Therapeutic Education: Psychological Support All cardiac transplant patients. On demand & scheduled Led by psychologists. Includes individual sessions, personality evaluation, and a support group (sometimes with a former transplant recipient).

Therapeutic Education: Transplant Info All cardiac transplant patients. Scheduled workshop "Understanding Your Cardiac Transplant," a workshop in small groups (3-5 patients) led by a clinician.

After the first CPET performed within the first week, the aerobic program consists of : i) a 30 (± 5) min MICT morning session at the power corresponding to the ventilatory threshold (PVT) ± 1 step, and monitored to correspond to a Borg-RPE 12-14 while progressing ; ii) a 24 to 36 min HIIT afternoon session, with 1 min interval at the power corresponding to the anaerobic threshold (PAT) ± 1 step, alternating with 3 min interval at ≤ 50% PVT, and monitored to correspond to a Borg-RPE ≥ 15 at the end of the session while progressing ; iii) All the other supplemental or non-aerobic exercises detailed in the general procedure.

When the AT is not reached/available during the first CPET, PVT +1 step is used initially and then adapted to the Borg-RPE scale.

A session is considered completed if 80% of the volume is made, at the targeted intensity.

Statistical analysis For the analysis, all patient data were reviewed exploratorily (exploratory database), but the primary "intention-to-treat" analysis was restricted to the "analytic database," comprising only patients who completed both admission and discharge CPETs (see Statistical Analysis section).

ELIGIBILITY:
Inclusion Criteria:

* De Novo Heart Transplant Recipients (HTR)

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: De novo HTR, after Heart failure from any etiology, at any age, from 3 University Transplantation units in the south-eastern quarter of France, admitted in our rehabilitation center for cardiac rehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 510 (Actual)
Dates: Start 2012-12-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
VO2peak | Baseline (Week 1) Discharge (Week 5)
  Main determinant of Exercise capacity, measured during a symptom-limited CardioPulmonary Exercise Test (CPET), performed in routine at our cardiac rehabilitation department

SECONDARY OUTCOMES:
VO2 vt/at | Baseline (Week 1) Discharge (Week 5)
  VO2 at the ventilatory threshold (VO2vt, ml/kg/min) VO2 at the anaerobic threshold (VO2at, ml/kg/min) during CPET
Heart rate | Baseline (Week 1) Discharge (Week 5)
  Peak Heart Rate (HRpeak, bpm) Heart rate at rest (HRrest, bpm) HR at VO2vt (HRvo2vt, bpm) HR at VO2at (HRvo2at, bpm) Heart Rate Reserve, i.e HRpeak-HRrest (HRR, bpm) during CPET
Power output | Baseline (Week 1) Discharge (Week 5)
  Maximum Work Power (Pmax, W) Work power at VT and AT (Pvt and Pat, W) during CPET
O2pulse | Baseline (Week 1) Discharge (Week 5)
  VO2peak / HRpeak ratio (ml/kg/min/bpm), during CPET
Echocardiography parameters | Baseline (Week 1) Discharge (Week 5)
  Ejection Fraction (%)
Biological Parameters/Renal Failure | Baseline (Week 1) Discharge (Week 5)
  eGFR by CKD-EPI (mL/min per 1.73 m2 ) Renal Failure: e.g None or Mild (eGFR ≥ 60 mL/min) Moderate (30 ≤ eGFR < 59.9 mL/min) Severe (15 ≤ eGFR ≤ 29.9 mL/min) Terminal (eGFR < 15 mL/min)
Clinical parameters | Baseline (Week 1)
  Sex (men)
Clinical Parameters | Baseline (Week 1)
  Age (year)
Clinical Parameters | Baseline (Week 1) Discharge 'Week 5)
  BMI (kg/m²)
Clinical Parameters | Baseline (Week 1) Discharge (Week 5)
  Graft - Rehabilitation Center admission time (day) Lenght of hospital-stay in Rehabilitation department (day)
Clinical Parameters | Baseline (Week 1) Discharge (Week 5)
  Etiology HF (%) (Dilated Cardiomyopathy- Ischaemic Cardiomyopathy- Congenital Cardiomyopathy- Hypertrophic Cardiomyopathy- Other Cardiomyopathy- ReGraft) ECMO (pre or post-HTx, %) Heartmate (%) Immunosuppressive medication (%) (Ciclosporine Tacrolimus Prednisolone)

IPD SHARING:
Plan to Share IPD: Undecided
Not enough time between end of data collection and open publication